CLINICAL TRIAL: NCT07347054
Title: Clinical Study of Myofascial Trigger Points(MTrPs) Injection in the Treatment of Chronic Musculoskeletal Pain(CMP), Chronic Migraine and Cervicogenic Headache
Brief Title: Clinical Study of Myofascial Trigger Points(MTrPs) Injection in the Treatment of Shoulder Osteoarthritis(OA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2025-317-02-03
Record Dates: First submitted 2025-12-27; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Myofascial Trigger Points; Chronic Musculoskeletal Pain; Shoulder Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint cavity injection group (Active Comparator): Joint cavity injection with triamcinolone acetonide.
  Interventions: Procedure: Joint Cavity Injection
- MTrPs injection group (Experimental): MTrPs injection with triamcinolone acetonide.
  Interventions: Procedure: MTrPs Injection

INTERVENTIONS:
Procedure: Joint Cavity Injection — Patients in the intra-articular injection group will receive an intra-articular shoulder injection via an anterolateral approach. The injection solution is prepared using 7 mL of 1% lidocaine and 1 mL of triamcinolone acetonide (40 mg/mL).
  Arms: Joint cavity injection group
Procedure: MTrPs Injection — The volume of infiltration solution is determined by the number of trigger points, with each trigger point receiving 1 mL of injection volume. The injection solution is prepared by combining 1 mL of triamcinolone acetonide (40 mg/mL), lidocaine, and normal saline, resulting in a final lidocaine concentration of 1%. A 25-gauge needle is used to inject perpendicular to the skin surface at the selected tender points, with the solution administered as a single bolus into each tender point within 10 seconds.
  Arms: MTrPs injection group

SUMMARY:
Chronic musculoskeletal pain (CMP) is a common disease in China, with a high incidence among the elderly, and has a significant impact on patients' quality of life. Shoulder osteoarthritis is a common type of CMP. Currently, both domestic and international studies have confirmed that glucocorticoid injection at myofascial trigger points(MTrPs) can alleviate patients' pain symptoms. MTrPs injection is safe and easy to operate, and can improve the clinical management efficiency of patients with shoulder osteoarthritis. Therefore, we designed a prospective, randomized controlled, blinded outcome, non-inferiority study to compare the long-term clinical efficacy of glucocorticoid injection at myofascial trigger points and complex intra-articular injection in treating shoulder osteoarthritis. Patients will be randomly divided into two groups and receive either glucocorticoid injection at MTrPs or joint cavities. After treatment, patients will be followed up for 2 years. Their NRS scores, WOMAC scores, Patient Global Impression of Change(PGIC) scale, and adverse reactions will be recorded at 2 weeks, 4 weeks, 8 weeks, 12 weeks, and 24 weeks. If the results indicate that the clinical efficacy of myofascial trigger point injection for shoulder osteoarthritis is not inferior to that of injection at intra-articular injection, it will provide a safe and simple treatment option that is easy to promote for patients who do not respond to conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of shoulder osteoarthritis with radiographic evidence of osteoarthritis (Kellgren-Lawrence grade 1-4) confirmed by at least two orthopedic surgeons, pain specialists, or general practitioners, with physical examination confirming at least one myofascial trigger point;
* Disease duration exceeding 3 months;
* Age ≥ 45 years;
* Numerical Rating Scale (NRS) score ≥ 3 points despite prior conservative pharmacological treatment;
* Signed informed consent form.

Exclusion Criteria:

* History of allergy to trial medications such as corticosteroids;
* Alcohol abuse; long-term use of opioids (exceeding 2 weeks or more than 3 days per week for over 1 month); suspected use of sedative or analgesic medications; patients on long-term steroid therapy;
* Severe neurological disorders, significant hepatic or renal dysfunction, heart failure, coagulation abnormalities, gastric ulcer, diabetes, inflammatory rheumatic diseases, etc.;
* Intra-articular injection within the past 6 months or planned joint replacement surgery;
* Inability to use pain assessment scales;
* Presence of local or systemic infection;
* Pregnant or lactating patients.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1036 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
NRS pain scores | at the 4-weeks
  The pain intensity of the shoulder will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.

SECONDARY OUTCOMES:
NRS pain scores | at the 2, 4, 8, 12, and 24 weeks
  The pain intensity of the shoudler will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
WOMAC scores | at the 2, 4, 8, 12, and 24 weeks
  The WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index) is a standardized instrument specifically designed to assess symptoms and function in patients with shoulder osteoarthritis. It comprises three dimensions with a total of 24 items: pain (5 items), stiffness (2 items), and physical function in daily activities (17 items). It utilizes a Likert scale (0-4 points, 0 = no symptoms), with a total score range of 0-96 points (or standardized to 0-100 points). Higher scores indicate greater functional impairment.
The Patient Global Impression of Change (PGIC) scale | at the 2, 4, 8, 12, and 24 weeks
  The Patient Global Impression of Change (PGIC) scale is a patient-rated instrument used to evaluate overall change in status following treatment. It employs a 7-point Likert scale (1 = "very much worse" to 7 = "very much improved"), focusing on the patient's subjective perception of symptoms, function, and quality of life. The evaluation criterion defines a score of 5 or higher as indicative of "improvement" (mild/moderate/marked), a score of 4 as "no change," and scores of 3 or below as "worsening."
Adverse Reactions | Through study completion, an average of 1 year
  Any systemic adverse reactions related to corticosteroids such as hyperglycemic reactions, infection at the puncture site, and intra-articular infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes